CLINICAL TRIAL: NCT00864825
Title: Allopurinol in Schizophrenia: A Randomized Trial Administering Allopurinol vs Placebo as add-on Antipsychotics in Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHEBA-09-6893-MW-CTIL
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Allopurinol; Add-on-treatment
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allopurinol (Experimental)
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator)
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Allopurinol — Allopurinol 1 capsule 300 mg, or placebo, bid (twice a day) for 42 days.
  Other Names: Alloril, Zylol, Zyloric

SUMMARY:
The objective of the study is to evaluate the efficacy of allopurinol, compared to placebo, as add-on to anti-psychotics in the treatment of patients with schizophrenia.

DETAILED DESCRIPTION:
An emerging body of evidence supports a purinergic hypothesis for schizophrenia. Adenosine agonists have been shown to have properties similar to those of dopamine antagonists and there is a well characterized antagonistic interaction between adenosine and dopamine receptors in the ventral striatum1. Increased adenosinergic transmission has been demonstrated to reduce the affinity of dopamine agonists for dopamine receptors. It has been theorized that adenosine may exert some of its antipsychotic effects through modulation of glutamatergic transmission.

Three double-blind, randomized, placebo-controlled trials have showed statistically significant greater improvements in PANSS scores in the allopurinol groups vs. placebo groups. These empiric data, together with the theoretical and basic science background cited, provide the impetus for this proposed study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-65 years of age, inclusive
2. Because gout is relatively rare in women of childbearing age, there are few reports describing the use of allopurinol during pregnancy; in those there were no adverse fetal outcomes attributable to allopurinol. Therefore, only females who are abstinent or practicing an established method of birth control (oral contraceptive tablets, hormonal implant device, hormone patch, injectable contraceptive, intrauterine device [IUD]) can be included in the trial.
3. Willing and able to provide informed consent, after the nature of the study has been fully explained
4. Current DSM-IV-TR diagnosis of schizophrenia as confirmed by SCID
5. Symptoms: 4 (moderate) or above on CGI-S AND >= 4 (moderate) score on two of the following four PANSS items: delusions, hallucinatory behaviors, conceptual disorganization or suspiciousness/ persecution.
6. Must be on any antipsychotic drug for at least 2 weeks prior to the baseline visit, at doses within the PORT criteria. Patients receiving higher doses will have their records reviewed to insure that dose is required. Patients receiving two anti-psychotics, or IM depot antipsychotics can also be included.
7. Inpatients or outpatients.

Exclusion Criteria:

1. Unwilling or unable, in the opinion of the Investigator, to comply with study instructions
2. Pregnant or breast-feeding
3. Unstable medical disease (malignancy, poorly controlled diabetes, active ischemic cardiac disease, or cardiomyopathy, serious pulmonary disease, , kidney disease, impaired liver functioning
4. Likely allergy or sensitivity to allopurinol
5. At significant risk of committing suicide, or in the opinion of the Investigator, currently is at imminent risk of suicide or harming others.
6. Suffers from a significant Substance Dependence disorder based on DSM-IV criteria within the 3 months prior to Screening, or is deemed by the Investigator to have a high risk of substance use during the study. Patients with a history of recreational use of cannabinoids or alcohol, and/or patients who smoke cigarettes can be included.
7. Concurrent delirium, mental retardation, drug-induced psychosis, or history of brain trauma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
PANSS total score. | 6 weeks

SECONDARY OUTCOMES:
PANSS positive, negative and general psychopathology scales, BACS, CGI, Simpson-Angus Scale. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Weiser, MD, Principal Investigator — Sheba Medical Center
Locations (33):
- Israel (10):
  - Abrabanel Mental Health Center, Bat Yam
  - Beer-Yaakov Mental Health Center, Beer-Yaakov
  - Shalvata Mental Health Center, Hod HaSharon
  - Jaffa Mental House Center, Jaffa
  - Herzog Medical Center, Psychiatry, Jerusalem
  - Kfar Shaul Mental Health Center, Jerusalem
  - Nes Ziona Mental Health Center, Ness Ziona
  - Shaar Menashe Mental Health Center, Shaar Menashe
  - Sheba Medical Center, Psychiatry Department, Tel Hashomer, Ramat Gan
  - Lev Hasharon Mental Health Center, Tsur Moshe
- Romania (23):
  - Spitalul Clinic de Urgenta Clinica "E. Pamfil" Timisoara, Bd. Iosif Bulbuca, 156, Jud Timis
  - Spitalul Clinic de Psihiatrie, sectia 14, Berceni St., 10-12, Bucharest
  - Spitalul Clinic de Psihiatrie, Clinica 9, Berceni St., 10-12, Sector 4, Bucharest
  - Spitalul Clinic de Psihiatrie, sectia 10, Berceni St., 10-12, Sector 4, Bucharest
  - Spitalul Clinic de Psihiatrie, sectia 12, Berceni St., 10-12, Sector 4, Bucharest
  - Spitalul clinic de Psihiatrie, sectia 13, Berceni St., 10-12, Sector 4, Bucharest
  - Spitalul Clinic de Psihiatrie, sectia 1, Berceni St., 10-12, Sector 4, Bucharest
  - Spitalul Clinic de Psihiatrie, sectia 3, Berceni St., 10-12, Sector 4, Bucharest
  - Spitalul Clinic de Psihiatrie, sectia 6, Berceni St., 10-12, Sector 4, Bucharest
  - Spitalul Clinic, sectia 8, Berceni St., Sector 4 Bucharest
  - Spitalul de Psihiatrie, Titan, Bld Nicolae Grigorescu, No. 41, Sector 3,
  - Spitalul Clinic de Urgenta Militar Sectia Psihiatrie Clinica, Bucuresti, Mircea Vulcanescu 88, Str. Vulcanescu, Nr. 88
  - Spitalul de Neuropsihiatrie Oradea, Cuza Voda St, 36, Oradea
  - Clinica de Psihiatrie nr.1, Gh. Marinescu St.38 ,Targu-Mures
  - Spitalul Clinic Judetean De Urgenta, Clinica Psihiatrie, Octavian Goga St, 17, Arad
  - Spitalul Clinic de Psihiatrie "Socola", Sos Bucium, 36, Iasi
  - Spitalul Clinic Colentina Cabinet Psihiatrie Ambulatoriu, Sos. Stefan Cel Mare Nr. 19-21, Sect. 2
  - Spitalul Clinic de Psihiatrie "Ghe. Preda", Str. Bagdazar 12, Sibiu
  - Spitalul Clinic Judetean de Urgenta -Cluj, Str. Clinicilor Nr. 3-5, 3400
  - Spitalul de Psihiatrie Botosani, Str. I.C.Bratianu Nr. 116, Botosani
  - Spitalul Clinic de Psihiatrie si Neurologie, Str. Prundului 7 - 9, Brasov
  - Spitalul Clinic Judetean, Sectia Clinica Psihiatrie, Str. Victor Babes, Nr. 43, Cluj Napoca
  - Spitalul de Psihiatrie si Neurologie, Str.Mihai Eminescu, Nr.18, Brasov

REFERENCES:
- [Derived] Weiser M, Gershon AA, Rubinstein K, Petcu C, Ladea M, Sima D, Podea D, Keefe RS, Davis JM. A randomized controlled trial of allopurinol vs. placebo added on to antipsychotics in patients with schizophrenia or schizoaffective disorder. Schizophr Res. 2012 Jun;138(1):35-8. doi: 10.1016/j.schres.2012.02.014. Epub 2012 Apr 4. PMID 22483162